CLINICAL TRIAL: NCT01906073
Title: An Open Label, Cross-over, Randomized Controlled Multicenter Phase III Study Comparing Standard Oral SR-morphine by the Clock Medications With Self-controlled Nasal Fentanyl for Chronic Cancer Pain Requiring Opioids
Brief Title: Nasal Fentanyl for Chronic Cancer Pain
Acronym: NFCP-2
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other); L'Hospitalet de Llobregat (Other); University Hospital, Bonn (Other); Cantonal Hospital of St. Gallen (Other); Maastricht University Medical Center (Other); Flinders University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NFCP-2
Record Dates: First submitted 2013-07-19; First posted 2013-07-23 (Estimated); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Cancer; Pain
Keywords: fentanyl; administration, intranasal; morphine; patient satisfaction; patient preference
MeSH Terms: conditions — Neoplasms; Pain; Patient Satisfaction; Patient Preference

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intranasal fentanyl spray (Experimental): Fentanyl for nasal administration (NF), is supplied as sprays containing a phosphate buffered solution of fentanyl citrate. NF is available in three strengths: 0.5 mg/ml, 1 mg/ml and 2 mg/ml in multiple-dose sprays. The corresponding doses are 50, 100 and 200 µg/puff. NF is applied as one puff in one nostril. One puff defines and equals one dose. Applying a puff to each nostril the upper dose can be increased to 400 µg. The doses used in this study are 50, 100, 200 ad 400µg. Fentanyl may be administered for up to 6 pain episodes/ 24 hours. For each pain episode, a dose of NF is self-administrated in one nostril. If pain relief is not achieved, another dose of NF could be administered in the opposite nostril after 15 minutes.
  Interventions: Drug: intranasal fentanyl spray
- slow release morphine (Active Comparator): The active substance is released gradually during its transit through the gastrointestinal tract. Slow release (SR) morphine is available in 5, 10, 30, 60, 100 and 200 mg. SR morphine is administered twice a day, usually every twelfth hour.
  Interventions: Drug: slow release morphine

INTERVENTIONS:
Drug: intranasal fentanyl spray
  Other Names: Instanyl
  Arms: intranasal fentanyl spray
Drug: slow release morphine
  Other Names: Morphine sulphate pentahydrate
  Arms: slow release morphine

SUMMARY:
Today, patients with cancer pain in need of opioids for moderate to severe pain get long-acting morphine twice a day and morphine tablets taken on demand in addition. This procedure might be based on the assumption that cancer pain is persistent, although the evidence to support whether this assumption applies to all cancer patients is lacking. Some cancer patients might not need a fixed dose of long-acting morphine.

Because of rapid pain relief, the new fentanyl drugs open for the possibility to take an opioid on demand when pain occurs.

A pilot study where 10 patients with cancer pain were treated with a rapid-acting fentanyl nasal spray taken on demand, showed that this treatment was apparently feasible and safe for these patients.

This approach is studied further in NFCP-II. The participants will be treated with rapid-acting fentanyl nasal spray and long-acting morphine in a crossover study. The primary outcome will be patient satisfaction.

The study will consist of a test dose of nasal fentanyl, a dose-finding phase and a treatment phase with either nasal fentanyl taken on demand or slow-released morphine taken twice a day. After 10 days of treatment there is a crossover and the opposite drug is used for the same participant. Morphine tablets can be taken on demand in all phases of the study.

The participants will meet the investigator at inclusion, at the crossover and at the end of treatment. During the study, a diary is filled in by the participants every morning. Questions about pain and side effects are answered. Satisfaction is measured at the crossover and at end of treatment while preference is measured at the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Cancer disease
2. Adult (older than 18 years)
3. Cancer-related pain > 4 on an 11 point Numerical Rating Scale (NRS)
4. In the need of opioids (step II or III)
5. Able to use nasal drugs.
6. Life expectancy of > 6 months
7. Karnofsky status > = 60
8. Women of child bearing potential must use adequate contraception
9. Informed consent given according to applicable requirements before any trial-related activities.

Exclusion Criteria:

1. Use of opioids for moderate and severe pain
2. History of substance abuse.*
3. Pathological conditions of the nasal cavity as contraindication to nasal fentanyl
4. Renal- or liver- failure, defined as creatinin > 150 and alanine-amino transferase (ALAT) > x 1.5 reference value
5. Sleep apnoea syndrome, severe chronic obstructive lung disease or illnesses leading to severe respiratory depression.
6. Psychiatric disease
7. Neurological disease giving dizziness or sedation
8. Cognitive impairment which makes the patient unable to complete questionnaires or not able to comply with the study procedures.
9. Previous or ongoing facial radiotherapy
10. Recurrent nose bleeding
11. Known hypersensitivity to the active substances or excipients of the study drugs
12. Pregnant or breastfeeding women
13. Treated with monoamine oxidase (MAO) inhibitor within the last 14 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
the difference in patient reported satisfaction between the two treatment sessions | 13 days
  measured by the Treatment Satisfaction Questionnaire for Medication (TSQM)

SECONDARY OUTCOMES:
Patient preference (overall; including pain relief, tolerance to adverse effects and convenience) of treatments after finishing the second part of the clinical study | 26 days
  5 point Likert scale
Overall rating of average pain control in the two treatment phases | 26 days
  measured by an 11- point numeric rating scale
Overall rating of average side effects in the two treatment phase | 26 days
  measured by an 11-point numeric rate scales

CONTACTS AND LOCATIONS:
Overall Officials: Stein Kaasa, MD prof, Study Director — Norwegian University of Science and Technology